CLINICAL TRIAL: NCT05872646
Title: The Effect of Cognitive Functions on Upper Extremity Functionality in Parkinson's Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Dudu ŞİMŞEK, MSc Physiotherapist, Pamukkale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PamukkaleU-sımsek-parkınson-01
Record Dates: First submitted 2023-03-10; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Parkinson; Cognitive Impairment; Upper Extremity Problem; Functional Disturbance
Keywords: Parkinson; Cognitive function; Upper extremity
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: patient and age-gender matched healthy groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient group (Experimental): parkınson patient group
  Interventions: Diagnostic Test: clinical assessment
- healthy group (Other): age-gender matched healthy group
  Interventions: Diagnostic Test: clinical assessment

INTERVENTIONS:
Diagnostic Test: clinical assessment — clinical staging
  Other Names: modifiye hoehn yahr

SUMMARY:
Parkinson's Disease (PD), first described by James Parkinson in 1817, is a progressive movement disorder that develops mainly as a result of the destruction of nigrostriatal dopaminergic neurons. The aim of our study is to determine the effect of cognitive functions on upper extremity functionality in individuals with Parkinson's Disease.

DETAILED DESCRIPTION:
Parkinson's Disease (PD), first described by James Parkinson in 1817, is a progressive movement disorder that develops mainly as a result of the destruction of nigrostriatal dopaminergic neurons. Involvement of nigrostriatal dopaminergic neurons is associated with the motor manifestations of the disease. The most common of these symptoms are; resting tremor, bradykinesia, rigidity and balance disorder. However, non-motor symptoms related to the involvement of nervous system structures other than the dopaminergic nigrostriatal system can be observed in PD. However, due to the predominance of motor symptoms in PD, it took many years to notice cognitive changes. Traditionally, cognitive impairments in PD have been expected to occur in the advanced stages of the disease. However, cognitive impairments in the early stages are reported in approximately 30-35% of patients. Cognitive dysfunction is defined in PD, ranging from mild impairments in certain cognitive domains to severe dementia. Cognitive impairment primarily affects executive and visuospatial functions, and memory is secondarily affected.

Executive functions are higher cognitive processes that use and modify information from many cortical sensory systems in the fore and hindbrain areas to modulate and teach behavior. The frontal cortex, especially the prefrontal cortex and its striatal connections are very important neuroanatomical regions for executive functions. The relationship between the effects of cognition and motor performance and parameters in groups such as the elderly, PD and Alzheimer's patients in which these centers are affected has been an issue that has attracted the attention of many researchers. Most of the studies have focused on the lower extremity performance of cognition. However , it has been reported that cognition has positive effects on upper extremity performance and early acquired upper extremity skills have positive effects on cognitive performance .

The aim of our study is to determine the effect of cognitive functions on upper extremity functionality in individuals with Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of Parkinson's Disease.
* Not having hearing and vision problems.
* To be able to take the commands required for the manual dexterity tests.
* Agree to participate in the study.

Exclusion Criteria:

* Having undergone musculoskeletal surgery for the upper extremity.
* Having vision and hearing problems.
* Having an additional disease that may affect cognitive tests.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Modified Hoehn Yahr Scale | 1 year
  Used for clinical staging of Parkinson's disease
Unified Parkinson's Disease Rating Scale | 1 year
  Used for the evaluation of clinical manifestations of Parkinson's disease
Parkinson's Disease Questionnaire-PDQ 39 | 1 year
  Used to assess the quality of life of Parkinson's patients

SECONDARY OUTCOMES:
Stroop Test | 1 year
  measures the selective attention ability of individuals
Wechsler Memory Scale-Revised | 1 year
  To assess attention, learning, memory and working memory in individuals aged 16-89
Dexterity Questionnaire-24 | 1 year
  To assess manuel dexterity
Nine Hole Peg Test | 1 year
  To assess manuel dexterity

CONTACTS AND LOCATIONS:
Overall Officials: DUDU ŞIMŞEK, Study Chair — PhD student
Locations (1):
- Pamukkale Unıversity, Denizli, Turkey (Türkiye)